CLINICAL TRIAL: NCT05348473
Title: Comparison of the Effects of Different Seton Application Techniques on the Quality of Life in the Postoperative Period in Perianal Fistula Disease
Brief Title: Changes in Patients' Quality of Life With Differences in Seton Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cihangir Akyol, Associate Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AUG-2021-0001
Record Dates: First submitted 2022-03-20; First posted 2022-04-27 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- alpha group (Active Comparator): In this group, tips of the seton will be tied as alpha-shaped
  Interventions: Device: Alpha type
- Beta group (Sham Comparator): The tips of the seton in this group will be overlapped and tied. There is no palpable free ends.
  Interventions: Device: Beta type
- Comfort group (Experimental): Knotless seton will be applied
  Interventions: Device: Comfort type

INTERVENTIONS:
Device: Alpha type — Tips of the seton will be tied as alpha-shaped.
  Arms: alpha group
Device: Beta type — Tips of the seton in this group will be overlapped and tied
  Arms: Beta group
Device: Comfort type — Knotless seton will be applied
  Arms: Comfort group

SUMMARY:
Investigators aim to investigate the changes in patients' quality of life with different type of seton application.

DETAILED DESCRIPTION:
Perianal fistula is a very common disease. Perianal fistula develops in the 50% of the anorectal abscess. Perianal fistulas are usually complications of recurrent anorectal abscesses. The management of the fistula is sometimes challenging and requires a long period of time. One of the treatment methods in perianal fistula is seton application. Seton is a rubber band made of various materials such as silicone, silk, latex, etc. It is passed through the fistula tract, and then the tips are tied to each other. Seton is usually kept there for 3 - 6 months depending on the condition of the fistula. Seton causes a foreign body reaction. After this process, there are various fistula management methods. Seton application is again one of the choices besides fistulotomy, fistulectomy, ablation methods, etc.

As seton is a frequently preferred method, patients should get used to living with seton. Severe irritation and a decrease in quality of life are observed in patients depending potentially on the seton binding methods.

Investigators aim to evaluate the seton application methods that will minimize the decrease in the quality of life in this difficult process for patients by comparing 3 different seton application methods that investigators apply in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* -Primary perianal fistula

Exclusion Criteria:

* Suprasphincteric fistula
* Patient who had previous perianal fistula surgery
* Crohn
* Radiotherapy
* Patient with pre-existing anal incontinence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-12-12 (Estimated); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life on 14th day | 14th day
  Quality of Life in patients with Anal Fistula Questionnaire (Qolaf-Q) will measure the quality of life in all groups. Minimum and maximum values are 17 and 85, respectively. Higher scores mean a worse outcome.
Quality of life on 30th day | 30th day
  Quality of Life in patients with Anal Fistula Questionnaire (Qolaf-Q) will measure the quality of life in all groups. Minimum and maximum values are 17 and 85, respectively. Higher scores mean a worse outcome.
Quality of life on 90th day | 90th day
  Quality of Life in patients with Anal Fistula Questionnaire (Qolaf-Q) will measure the quality of life in all groups. Minimum and maximum values are 17 and 85, respectively. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet A Koç, MD, Study Director — Ankara Üniversitesi Tıp Fakültesi
Locations (1):
- Ankara University School of Medicine Department of General Surgery, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrer-Marquez M, Espinola-Cortes N, Reina-Duarte A, Granero-Molina J, Fernandez-Sola C, Hernandez-Padilla JM. Analysis and description of disease-specific quality of life in patients with anal fistula. Cir Esp (Engl Ed). 2018 Apr;96(4):213-220. doi: 10.1016/j.ciresp.2017.12.003. Epub 2018 Feb 13. English, Spanish. PMID 29452968
- [Background] Kristo I, Stift A, Staud C, Kainz A, Bachleitner-Hofmann T, Chitsabesan P, Riss S. The type of loose seton for complex anal fistula is essential to improve perianal comfort and quality of life. Colorectal Dis. 2016 Jun;18(6):O194-8. doi: 10.1111/codi.13335. PMID 26999764
- [Background] Ferrer-Marquez M, Espinola-Cortes N, Reina-Duarte A, Granero-Molina J, Fernandez-Sola C, Hernandez-Padilla JM. Design and Psychometric Evaluation of the Quality of Life in Patients With Anal Fistula Questionnaire. Dis Colon Rectum. 2017 Oct;60(10):1083-1091. doi: 10.1097/DCR.0000000000000877. PMID 28891853
- [Derived] Ozgu K, Kutlu B, Koc MA, Ersoz S, Gokmen D, Akyol C. Assessing quality of life in anal fistula patients after Seton placement using different knot types: Randomized controlled trial. Int J Colorectal Dis. 2026 Jan 29;41(1):52. doi: 10.1007/s00384-026-05099-6. PMID 41612009
- See also: Análisis y descripción de la calidad de vida específica en pacientes con fístula analAnalysis and description of disease-specific quality of life in patients with anal fistula — https://doi.org/10.1016/j.ciresp.2017.12.003